CLINICAL TRIAL: NCT06111027
Title: Usability of Laryngeal Vibro-tactile Stimulation as a Non-invasive Treatment for the Voice Disorder Spasmodic Dysphonia
Brief Title: Usability of Vibro-tactile Stimulation to Treat Spasmodic Dysphonia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00019659
Record Dates: First submitted 2023-10-16; First posted 2023-11-01 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Spasmodic Dysphonia; Laryngeal Dystonia
MeSH Terms: conditions — Dysphonia

STUDY DESIGN:
Intervention Model Description: Usability study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Will use the device, single group
  Interventions: Device: Vibro-tactile stimulation

INTERVENTIONS:
Device: Vibro-tactile stimulation — Vibro-tactile stimulation is a non-invasive treatment option. As stimulators, we will apply a pair of light-weight encapsulated cylindrical vibrators to both sides of the larynx (voice box). The vibration frequency for VTS will set be to 100Hz and the participant may feel a mild tingling or vibrating sensation during VTS. The participants will be asked to apply for VTS at home over a period of 8 weeks. The participants will be asked to use this device for 3 days in the first week, 4 days in the second week, 5 days in the third week and 6 days in the fourth week. During the last 4 weeks, the participants will apply VTS on self-selected days as needed, not exceeding 6 times a week, to control and improve symptoms.

SUMMARY:
The general aim of the study is to provide evidence for usability and feasibility of applying vibro-tactile stimulation (VTS) at home as a non-invasive form of neuromodulation to improve speech in people with spasmodic dysphonia (SD). This work addresses a clinical need to develop alternative or auxiliary treatments for a rare voice disorder with very limited treatment options. Successful completion of the proposed work will be an important step in advancing laryngeal VTS as a therapeutic intervention for improving voice symptoms in SD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of spasmodic dysphonia (laryngeal dystonia) for a minimum of 6 months with documented symptom relief after Botox injection.
* Diagnosis is made by a voice disorder specialist.

Exclusion Criteria:

* Regular intake of benzodiazepines
* Cognitive impairment: score < 27 on Mini-mental state examination
* Identifies with a neurological or musculoskeletal impairment affecting speech motor function. These impairments may include a form of: Dyskinesia, Dystonia, Essential Tremor, Huntington's Disease, Multiple System Atrophy, Muscle Tension Dysphonia, Parkinsonism, Progressive Supranuclear Palsy, Spasticity, Intracranial Neoplasm (brain tumor), Spinal Neoplasm, Cerebrovascular Accident (Stroke), Mild Traumatic Brain Injury, Intracranial Hemorrhage, Multiple Sclerosis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Perceived voice effort | 8 weeks
  Participants will rate their perceived effort level of vocalization on an ordinal scale of 0 to 10 (0 being with no effort and 10 being with maximal effort). The recordings will provide subjective impression of treatment.

SECONDARY OUTCOMES:
The number of voice breaks | 8 weeks
  Prior to study begin, participants will receive a manual with instructions about the remote audio recording procedure. During pre- and post-application assessment, participants will record their voices using a voice recording application on their smartphone or digital tablet. The recordings will provide objective data on the number of voice breaks.
The duration of voice break | 8 weeks
  Prior to study begin, participants will receive a manual with instructions about the remote audio recording procedure. During pre- and post-application assessment, participants will record their voices using a voice recording application on their smartphone or digital tablet. The recordings will provide objective data on the duration of voice breaks.

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Konczak, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States